CLINICAL TRIAL: NCT06123585
Title: Artificial Intelligence (AI) Empowered Smile Simulations: Do They Accurately Predict Actual Post Treatment Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: SRB/SDC/ORTHO-2119/23/019
Record Dates: First submitted 2023-11-01; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Invisalign® SmileView™ (Experimental)
  Interventions: Other: Invisalign® SmileView™
- Invisalign aligners (Active Comparator)
  Interventions: Other: Invisalign aligners

INTERVENTIONS:
Other: Invisalign® SmileView™ — Pretreatment smiles were captured using the Invisalign® SmileView™ to simulate their new smiles before treatment was started.
  Arms: Invisalign® SmileView™
Other: Invisalign aligners — Patients were then treated using upper and lower Invisalign aligners with average treatment time of 12±3 months.
  Arms: Invisalign aligners

SUMMARY:
The aim of the present study is to assess the predictability of Invisalign® SmileView™ for digital AI smile simulation in comparison to actual smile treatment outcomes, using various smile assessment parameters.

ELIGIBILITY:
Inclusion Criteria:

* healthy systemic condition with no chronic diseases
* no previous orthodontic treatment
* adequate oral hygiene
* a healthy periodontium.

Exclusion Criteria:

* chronic diseases
* previous orthodontic treatment
* poor oral hygiene
* periodontal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-05 (Actual)

PRIMARY OUTCOMES:
Smile line | through study completion, an average of 1 year
  The extent of the vertical tooth display on smiling or the elevation of the upper lip in relation to the maxillary incisors. Three types of smile lines have been described- high, average, and low. A high smile shows the maxillary anterior teeth along with a significant amount of gingiva, an average smile shows maxillary anterior teeth with only interproximal gingiva, and a low smile typically shows less than two-thirds of the maxillary anterior teeth
Smile arc | through study completion, an average of 1 year
  The relationship between the curvature of the maxillary anterior teeth and upper border of the lower lip. It is defined by drawing a line along the maxillary central incisal edges to the cusp tips of maxillary canines, which is related to another line drawn across the superior border of the lower lip. In subjects whose maxillary teeth are covered by lower lip, smile arc is designated as "not available". Three types of smile arcs have been described- "parallel to the teeth" (when the two lines follow the same curvature) also called a consonant smile, and a non-consonant smile, if the two lines are not parallel. A non-consonant smile can either be "straight" (with flatter curvature of the maxillary anterior teeth in relation to the lower lip) or "reverse" (when the maxillary anterior teeth form a reverse curve in relation to lower lip).
The most posterior teeth displayed | through study completion, an average of 1 year
  Smiles are categorized as displaying teeth up to the canines, first premolars, second premolars, or the first molars. A tooth is counted when more than half of its surface is visible.
The philtrum height | through study completion, an average of 1 year
  Distance measured in millimeters from subspinale (the base of the nose at the midline) to the most inferior portion of the upper lip on the vermilion tip beneath the philtral columns
Commissure height | through study completion, an average of 1 year
  Distance measured in millimeters from a line constructed from the alar bases through subspinale and then from the commissures perpendicular to this line. The differential lip growth exhibits the difference in height in philtrum and commissural height in adolescents.
Smile width/Inter-commissure width | through study completion, an average of 1 year
  The distance (mm) from outer commissure to outer commissure on smile in millimeters.
Smile index | through study completion, an average of 1 year
  The ratio between the horizontal smile width and the vertical smile height during smiling (smile width/smile height).
Maxillary inter-canine width | through study completion, an average of 1 year
  distance from the distal aspect of the right canine to the distal aspect of the left canine in millimeters
Buccal corridor | through study completion, an average of 1 year
  It is the space created between the buccal surface of the posterior teeth and the lip corners when the patient smiles. Orthodontists often refer to buccal corridors as "negative spaces". The buccal corridor is measured from the mesial line angle of the maxillary first premolars to the interior portion of the commissure of the lips. Moore et al [16]. have previously quantified a buccal corridor of 28% as medium-narrow, 15% as medium, 10% as medium-broad, and 2% as broad smile fullness
Amount of lower incisor show | through study completion, an average of 1 year
  The amount of lower incisor display which can be categorized into either 1) No show of lower incisors during smiling, 2) partial lower incisor exposure or 3) full length lower incisor exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Samar M Adel, PhD, Principal Investigator — Alexandria University; Yashodhan M Bichu, DSATP, Study Chair — Faculty of Dentistry, University of British Columbia, Vancouver, Canada; Srirengalakshmi Muthuswamy Pandian, PhD, Study Chair — Saveetha Dental College, Saveetha Insitute of Medical and Technical Sciences, Chennai, India.; Waddah Sabouni, Study Chair — Private Practice, Invisalign Centre Dubai United Arab Emirates.; Chandani Shah, Study Chair — Private practice, Mumbai, India; Nikhillesh Vaid, PhD, Study Chair — Saveetha Dental College, Saveetha Insitute of Medical and Technical Sciences, Chennai, India.
Locations (1):
- Private orthodontic offices of Invisalign Diamond Plus Elite, Dubai, United Arab Emirates

REFERENCES:
- [Derived] Adel SM, Bichu YM, Pandian SM, Sabouni W, Shah C, Vaiid N. Clinical audit of an artificial intelligence (AI) empowered smile simulation system: a prospective clinical trial. Sci Rep. 2024 Aug 21;14(1):19385. doi: 10.1038/s41598-024-69314-6. PMID 39169095